CLINICAL TRIAL: NCT02329236
Title: Prevalence of Attention Deficit Disorder Among Patients With Constitutional Growth Delay
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dror Nitsan, medical doctor, Meir Medical Center
Other Study IDs: meir medical center
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Attention-deficit/Hyperactivity Disorder; Constitutional Growth Delay
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Puberty, Delayed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- children with constitutional growth delay
- children with Familial short stature

SUMMARY:
The aim of the our study is to investigate whether there is an increased incidence of ADHD ( based on self reports and questionnaires) among children with short stature due to constitutional growth delay (CGD) in comparison with children with Familial short stature.

DETAILED DESCRIPTION:
Filling out the study questionnaire by ADHD diagnosed and suspected children (have a positive DBDRS (Disruptive Behavior Disorders Rating Scale Questionnaire) result) who were referred to the pediatric endocrine clinic of our hospital for short statue evaluation. The study questionnaire will be filled by child's guardian.

The study and the DBDRS questionnaires will be filled only after obtaining an informed consent.

The required data including growth statistics, age at puberty, bone age and other relevant data will be collected from the child's medical records.

The data on patients will be processed anonymously.

ELIGIBILITY:
Inclusion Criteria:

* undergo evaluation and follow-up due to short stature caused by either CGD or Familial short stature

Exclusion Criteria:

* Children with short stature due to other reasons such as hormonal disorders (thyroid disorders, growth hormone deficiency), genetic syndromes

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with short stature due to constitutional growth delay or familial short stature followed at the endocrine unit.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
incidence of ADHD among children with short stature due to constitutional growth delay (CGD) in comparison with children with Familial short stature | single point in time during the visit at the endocrine clinic